CLINICAL TRIAL: NCT07402707
Title: Dosing of Steroids for Acute Asthma Given in the Emergency Department - a Pilot Randomised Feasibility Trial of Dexamethasone in Children
Acronym: DOSAGE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCH- 2695
Record Dates: First submitted 2025-02-18; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Acute Asthma; Dexamethasone
Keywords: Dexamethasone
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.3mg dose (Other): Lower dose of dexamethasone
  Interventions: Drug: dexamethasone oral
- 0.6mg (Other): Lower dose of dexamethasone
  Interventions: Drug: dexamethasone oral

INTERVENTIONS:
Drug: dexamethasone oral — The interventions are Dexamethasone, 0.3mg/kg versus 0.6 mg/kg

SUMMARY:
Steroids given by mouth are an important first line treatment for children presenting with asthma attacks. Dexamethasone is the steroid used in some emergency departments (EDs) because of the need for a single dose and as it is well tolerated. The dose of dexamethasone in treating asthma attacks is not clearly established. This study compares two different doses of dexamethasone in children presenting with an asthma attack. Investigators will compare the effect of two different doses in reducing the need for a repeat prescription of steroids for an asthma attack in the 2 weeks after the first treatment. The investigators will also look at how often children attend the ED or their GP after being given treatment as well as the acceptability to parents and children. Although this study may provide an answer to the question of whether the different doses have the same effect, the investigators believe that a larger study will be needed to provide robust generalisable evidence, as well as to ensure that the outcomes are truly what matters to parents, children and healthcare professionals. This study will provide valuable information to enable a larger study to be undertaken.

DETAILED DESCRIPTION:
Asthma is the most common chronic condition to affect children, with approximately 1.1 million children treated for asthma in the UK. Hospital episode statistics confirm that emergency department (ED) attendances for exacerbations of asthma have risen over the past year, and accounts for a significant number of ED attendances and hospital admissions. Nearly 1000 children attended the ED at Sheffield Children's Hospital for asthma in 2022-23, with almost half requiring admission.

Steroids/glucocorticoids are first line treatments for acute exacerbations of asthma. The anti-inflammatory action of steroids reduces the airway oedema and secretions associated with acute asthma exacerbations, and their effects may be noted within two to four hours of administration. Traditionally, oral prednisolone has been the treatment used most widely. Prednisolone given orally is often vomited by the child and needs to be taken for 3-5 days. Dexamethasone is an alternative steroid which is better tolerated and due to its long duration of action can be used as a single dose given in the ED. Studies comparing prednisolone and Dexamethasone have demonstrated that Dexamethasone is non-inferior to Prednisolone in the treatment of asthma exacerbations (1,2). A systematic review found no differences between the two steroids in terms of hospital admission rates, time spent in the ED or relapse events, however children receiving Dexamethasone experienced lower noncompliance and vomiting rates. (3) Practically, use of dexamethasone allows simplification of treatment in EDs and improves flow as children do not have to wait for discharge medication. Treatment with Dexamethasone is more cost effective and treatment adherence is better.

In a survey of 37 UK EDs undertaken by the study team, 19 departments currently use Prednisolone, and 18 use Dexamethasone. Of the latter, 7 use 600 micrograms/kg and the other 11 use 300 micrograms/kg. The currently used dose at our institution is 600 micrograms/kg. The dose of dexamethasone used as oral treatment for exacerbations of asthma is not well established, as demonstrated by the survey and this reflects the studies which sought to compare Prednisolone with Dexamethasone which used different doses and routes. (4-6) While systemic steroids are an effective and safe treatment, there is a dose-dependent profile of side effects, hence the lowest effective dose should be used. This is even more important given concerns over side effects from even shorter courses of steroids as used in asthma (7). Dexamethasone is well established in the treatment of other acute paediatric respiratory conditions, such as croup, with evidence demonstrating that lower doses (150micrograms/kg) are safer, and equally as effective as higher doses (600 micrograms/kg) in this condition. (8, 9) The investigators hypothesise that using a lower dose of Dexamethasone (300 micrograms/kg) is not inferior to the 600 microgram/kg dose in the treatment of acute asthma. The effectiveness of treatment can be measured as length of stay in hospital or time to improvement in respiratory distress severity scores, however both of these can be subjective. Need for re-treatment with steroids is a pragmatic surrogate of efficacy of treatments as well as the need for further unscheduled medical care in children with asthma exacerbations. In our patient and parent involvement work for this study, parents have agreed that this outcome is important. They also want to be reassured that an effective dose is being given but are supportive of the study's objective and think it an important research question.

The investigators hypothesise that children treated with either dose of dexamethasone have a similar rate of retreatment with oral steroids (dexamethasone or prednisolone) for their asthma exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-15 years (inclusive) presenting to the ED with an asthma exacerbation, where oral steroids are recommended by Trust/National guidelines.
* Children whose parents/carers do not speak English will also be eligible provided they speak one of the common languages where an interpreter and Information Sheets are available (Slovakian, Arabic and Urdu).

Exclusion Criteria:

* Children who have been treated with oral or IV steroids in the last 2 weeks.
* Hypersensitivity to the study drug.
* Children who have concomitant stridor.
* First episode of wheezing (not previously diagnosed as asthma).
* Children with known difficult asthma who receive longer courses of steroids as standard.
* Life threatening episode of asthma.
* Children with other conditions that require them to have steroids when unwell.
* Children who are involved in current research or have recently been involved in research prior to recruitment

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Participant recruitment | 7 months
  The primary outcomes will be recruitment rate and time, attrition, willingness to be randomised, completion and follow-up rates

SECONDARY OUTCOMES:
Tolerability | 7 months
  Secondary outcomes of tolerability, mean abbreviated Asthma Control Test (ACT)
Tolerability | 7 months
  Asthma Control Questionnaire (ACQ) scores,
Tolerability | 7 months
  Reliever (Salbutamol) use
Tolerability | 7 months
  Need for repeat steroid prescription
Hospital Admission | 7 months
  Hospital admission, length of stay and unscheduled return visits to a health care practitioner within 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Gilchrist, Principal Investigator — Sheffield Children's NHS Foundation Trust
Locations (1):
- Sheffield Children's NHS Foundation Trust, Sheffield, United Kingdom